CLINICAL TRIAL: NCT00001044
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled HIV-1 Vaccine Trial to Evaluate the Safety and Immunogenicity of rgp120/HIV-1MN (Genentech) in Combination With QS21 Adjuvant and/or Alum in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 016; 10564 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Drug Therapy, Combination; Adjuvants, Immunologic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Aluminum Hydroxide; saponin QA-21V1

INTERVENTIONS:
Biological: Aluminum hydroxide
Biological: QS-21
Biological: rgp120/HIV-1MN

SUMMARY:
PRIMARY: To examine the safety and potential improvement in immune responses elicited by combining rsgp120/HIV-1MN with the adjuvant QS-21. SECONDARY: To examine the role of alum in the vaccine/adjuvant formulation; to determine the optimal dose ratio of vaccine to adjuvant; and to obtain initial information on the optimal schedule of administration. AS PER AMENDMENT 07/02/97: To determine the ability of immunization with rsgp120/HV-1MN in combination with QS21 with or without alum to induce an HIV-1 envelope-specific delayed-type hypersensitivity (DTH) response in volunteers who undergo rsgp120/MN skin testing.

Immune responses in HIV-uninfected individuals receiving subunit envelope vaccines formulated with alum adjuvant suggest that functional antibodies capable of neutralizing HIV-1 in vitro may be induced, but the titers are relatively low in comparison to those measured in individuals with natural HIV-1 infection. These limitations might be overcome by the addition or substitution of a more suitable adjuvant such as QS-21.

DETAILED DESCRIPTION:
Immune responses in HIV-uninfected individuals receiving subunit envelope vaccines formulated with alum adjuvant suggest that functional antibodies capable of neutralizing HIV-1 in vitro may be induced, but the titers are relatively low in comparison to those measured in individuals with natural HIV-1 infection. These limitations might be overcome by the addition or substitution of a more suitable adjuvant such as QS-21.

Volunteers are randomized to 20 treatment arms containing four patients each. rsgp120/HIV-1MN is administered at four dose levels: 0, 100, 300, and 600 mcg, and QS-21 adjuvant is administered at three dose levels: 0, 50, and 100 mcg. Some subject cohorts receive alum in the vaccine formulation. Sixty volunteers receive injections at months 0, 1, and 10, and 20 volunteers receive injections at months 0, 1, and 6. AS PER AMENDMENT 07/02/97: All consenting volunteers who have received three immunizations will be tested for DTH response to HIV-1 envelope with use of intradermal MN rsgp120. Follow-up is extended to 56 days after administration of the intradermal injections.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* HIV negativity by ELISA within 6 weeks of immunization.
* CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Hepatitis B surface antigen.
* Medical or psychiatric condition or occupational responsibilities that preclude compliance.
* Active syphilis. NOTE: Subjects with serology documented to be false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of allergy to thimerosal.
* AS PER AMENDMENT 07/02/97: History of eczema or allergic-type reactions to rsgp120/HIV-1MN vaccine (for volunteers undergoing DTH testing).

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. (NOTE: Medically indicated subunit or killed vaccines, such as influenza or pneumococcal, are allowed but should be given at least 2 weeks prior to HIV immunizations.)
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.
* AS PER AMENDMENT 07/02/97: Use of systemic steroids in the past month (for volunteers undergoing DTH testing).

Prior Treatment:

Excluded:

* Receipt of blood products or immunoglobulin within the past 6 months.

Identifiable high-risk behavior for HIV infection as determined by screening questionnaire, including history of injection drug use within the past year and higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Study Completion 1995-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McElrath J, Study Chair
Locations (4):
- United States (4):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - JHU AVEG, Pittsburgh, Pennsylvania
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Evans TG, McElrath MJ, Matthews T, Montefiori D, Weinhold K, Wolff M, Keefer MC, Kallas EG, Corey L, Gorse GJ, Belshe R, Graham BS, Spearman PW, Schwartz D, Mulligan MJ, Goepfert P, Fast P, Berman P, Powell M, Francis D; NIAID AIDS Vaccine Evaluation Group. QS-21 promotes an adjuvant effect allowing for reduced antigen dose during HIV-1 envelope subunit immunization in humans. Vaccine. 2001 Feb 28;19(15-16):2080-91. doi: 10.1016/s0264-410x(00)00415-1. PMID 11228380
- [Background] Zolla-Pazner S, Alving C, Belshe R, Berman P, Burda S, Chigurupati P, Clements ML, Duliege AM, Excler JL, Hioe C, Kahn J, McElrath MJ, Sharpe S, Sinangil F, Steimer K, Walker MC, Wassef N, Xu S. Neutralization of a clade B primary isolate by sera from human immunodeficiency virus-uninfected recipients of candidate AIDS vaccines. J Infect Dis. 1997 Apr;175(4):764-74. doi: 10.1086/513969. PMID 9086128